CLINICAL TRIAL: NCT01574807
Title: A Prospective, Randomized, Double-blind Study of the Anesthetic Efficacy of 3% Mepivacaine Plus 2% Lidocaine With 1:100,000 Epinephrine for Inferior Alveolar Nerve Blocks.
Brief Title: The Anesthetic Efficacy of 3% Mepivacaine Plus 2% Lidocaine With 1:100,000 Epinephrine for Lower Jaw Dental Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Nusstein, Associate Professor and Chair, Divison of Endodontics, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Endo-Lam2012
Record Dates: First submitted 2012-04-02; First posted 2012-04-10 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: mepivacaine; lidocaine; inferior alveolar nerve block; pulpal anesthesia; mepivacaine/lidocaine; lidocaine/lidocaine
MeSH Terms: conditions — Pain | interventions — Mepivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mepivacaine + lidocaine followed by lidocaine + lidocaine (Experimental): A repeated measures design utilizing a single group of subjects was employed with each subject serving as his/her own control. Each subject received two interventions: 1.) 1.8 cc 3% mepivacaine and 1.8 cc 2% lidocaine with 1:100,000 epinephrine (3% mepivacaine/2% lidocaine with epinephrine - combination 1) and 2.) 1.8 cc 2% lidocaine with 1:100,000 epinephrine followed by 1.8 cc 2% liocaine with 1:100,000 epinephrine at two seperate appointments spaced 2 weeks apart.
  Interventions: Drug: mepivacaine + lidocaine followed by lidocaine +lidocaine
- lidocaine + lidocaine followed by mepivacaine plus lidocaine (Experimental): A repeated measures design utilizing a single group of subjects was employed with each subject serving as his/her own control. Each subject received two interventions: 1.) 1.8 cc 2% lidocaine with 1:100,000 epinephrine and 1.8 cc 2% lidocaine with 1:100,000 epinephrine and 2.) 1.8 cc 3% mepivacaine and 1.8 cc 2% lidocaine with 1:100,000 epinephrine followed by 1.8 cc 2% liocaine with 1:100,000 epinephrine at two separate appointments spaced two weeks apart.
  Interventions: Drug: lidocaine + lidocaine followed by mepivacaine + lidocaine

INTERVENTIONS:
Drug: mepivacaine + lidocaine followed by lidocaine +lidocaine — 1.8 mL of 3% mepivacaine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine
  Other Names: Combo 1
  Arms: mepivacaine + lidocaine followed by lidocaine + lidocaine
Drug: lidocaine + lidocaine followed by mepivacaine + lidocaine — 1.8 mL of 2% lidocaine with 1:100,000 epinephrine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine followed by 1.8 mL of 3% mepivacaine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine
  Other Names: Combo 2
  Arms: lidocaine + lidocaine followed by mepivacaine plus lidocaine

SUMMARY:
The inferior alveolar nerve block (shot) is the most frequently used injection technique for achieving local anesthesia (numbness) for the teeth in the lower jaw. However, this injection does not always result in successful pulpal (tooth) anesthesia (patient felt pain). No study has combined mepivacaine and lidocaine anesthetics (numbing solutions) for this type of injection (shot). The investigators propose to compare an injection of mepivacaine followed by lidocaine to an injection of lidocaine followed by lidocaine to determine if there is a difference in effectiveness.

DETAILED DESCRIPTION:
One hundred adult male and female subjects will randomly receive two sets of inferior alveolar block injections (shots) consisting of; 1.) an injection of 1.8 mL of 3% mepivacaine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine, and 2.) an injection of 1.8 mL of 2% lidocaine with 1:100,000 epinephrine followed by 1.8 mL of 2% lidocaine with 1:100,000 epinephrine, at two separate appointments spaced at least two weeks apart, in a crossover design. Whether the subject receives the mepivacaine or the lidocaine for the first injection will be determined randomly. The doctor will not know whether the subject receives mepivacaine or lidocaine for the first injection. The subject will not know which anesthetics he/she receives. A pulp tester will be used to test the lower jaw teeth (molars, premolars, and incisors) for anesthesia (numbness) in 4-minute time cycles for 60 minutes. The data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65 years
* good health (ASA classification I or II)
* able to provide informed consent

Exclusion Criteria:

* allergy to lidocaine or mepivacaine
* history of significant medical problem (ASA classification III or greater)
* depression
* have taken CNS depressants (including alcohol or any analgesic medications) within the last 48 hours
* lactating or pregnant
* inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nusstein, DDS, MS, Principal Investigator — Chair, Division of Endodontics
Locations (1):
- The Ohio State University College of Dentistry, Postle Hall, Columbus, Ohio, United States

REFERENCES:
- [Background] Nusstein J, Reader A, Beck FM. Anesthetic efficacy of different volumes of lidocaine with epinephrine for inferior alveolar nerve blocks. Gen Dent. 2002 Jul-Aug;50(4):372-5; quiz 376-7. PMID 12640855
- [Background] McLean C, Reader A, Beck M, Meryers WJ. An evaluation of 4% prilocaine and 3% mepivacaine compared with 2% lidocaine (1:100,000 epinephrine) for inferior alveolar nerve block. J Endod. 1993 Mar;19(3):146-50. doi: 10.1016/s0099-2399(06)80510-8. PMID 8509754
- [Background] Cohen HP, Cha BY, Spangberg LS. Endodontic anesthesia in mandibular molars: a clinical study. J Endod. 1993 Jul;19(7):370-3. doi: 10.1016/S0099-2399(06)81366-X. PMID 8245762
- [Background] Rood JP, Caruana PE, Danford M, Pateromichelakis S. Prilocaine -- an investigation into its use in the presence of inflammation and in combination with lignocaine. J Dent. 1981 Sep;9(3):240-7. doi: 10.1016/0300-5712(81)90061-0. No abstract available. PMID 7024357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from august 2011 to May 2013 in the dental clinic of the College of Dentistry.
Pre-assignment Details: No subjects were excluded from the study.
Groups:
- Mepi/Lido + Lido/Lido Group: This group received Mepivacaine + lidocaine at 1st appointment and lidocaine + lidocaine at 2nd appointment.
- Lido/Lido + Mepi/Lido Group: This group received injections of lidocaine + lidocaine at 1st appointment and Mepivacaine + lidocaine at second appointment.
Period: First Appointment
Arm/Group | Mepi/Lido + Lido/Lido Group | Lido/Lido + Mepi/Lido Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Wash Out Period 2 Weeks
Arm/Group | Mepi/Lido + Lido/Lido Group | Lido/Lido + Mepi/Lido Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Second Appointment
Arm/Group | Mepi/Lido + Lido/Lido Group | Lido/Lido + Mepi/Lido Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants receive 3% mepivacaine + 2% lidocaine versus 2% lidocaine + 2% lidocaine injections in different randomized sequences.
Arm/Group | All Participants
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Pulpal Anesthesia Success.
Description: An electric pulp tester will be used to test the lower jaw teeth (molars, premolars, and incisors) for anesthesia (numbness) in 4-minute time cycles for 60 minutes. Measurements of less than 80 on the EPT is considered not numb (anesthesia failure). Readings of 80 equate to anesthetic success.
Time Frame: 60 minutes per injection sequence.
Population: Success of anesthesia was determined by subject achieving maximal level (80) with testing device by 5th testing time period (17 min.) following injection and maintaining that maximal response for the remainder of the testing time.
Measure: Count of Participants; unit: Participants
Groups:
- Mepivacaine + Lidocaine: Clinical appointment where: 1.8cc 3% mepivacine + 1.8cc 2% lidocaine is injected.
- Lidocaine + Lidocaine: Clinical appointment where - 1.8cc 2% lidocaine + 1.8cc 2% lidocaine is injected.
Arm/Group | Mepivacaine + Lidocaine | Lidocaine + Lidocaine
Number analyzed (Participants) | 100 | 100
Participants | 44 | 40
Statistical Analysis 1: Comparison: Mepivacaine + Lidocaine vs Lidocaine + Lidocaine; Test type: Superiority; p = 1.00, McNemar — Multiple McNemar tests corrected with Step-down Bonferroni method of Holm. A priori threshold for significance was 0.05; Percentage difference = 0

ADVERSE EVENTS:
Groups:
- Treatment Group: 3% mepivacaine/2% lidocaine with epinephrine - combination 1
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No